CLINICAL TRIAL: NCT07007585
Title: Risk Factors for Hospitalization and Transfusion Criteria in Patients With Dengue Virus Infection: A Prospective Observational Study
Brief Title: Risk Factors for Hospitalization and Transfusion Criteria in Patients With Dengue Virus Infection
Acronym: DENGUE-FACT
Status: Recruiting | Type: Observational
Sponsor: Jose Ivan Rodriguez de Molina Serrano (Other)
Responsible Party: Sponsor-Investigator, Jose Ivan Rodriguez de Molina Serrano, Head of Research and Medical Education Clinica Mexico, Clinica Mexico
Organization: Clinica Mexico (Other)
Other Study IDs: CMX0003
Record Dates: First submitted 2025-05-27; First posted 2025-06-06 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Dengue; Dengue Fever; Dengue Fever With Warning Signs
Keywords: Dengue; Hospitalization; Transfusion; Hemorrhagic Fever; Thrombocytopenia; Mexico
MeSH Terms: conditions — Dengue; Hemorrhagic Fevers, Viral; Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Inpatient Confirmed Dengue Cohort: This cohort includes patients aged 5 years and older with laboratory-confirmed dengue virus infection (via NS1 antigen, IgM serology, or PCR) who present to the emergency department or outpatient clinic at Clínica México. Patients are prospectively followed from initial presentation through resolution of illness or hospital discharge. No interventions are administered as part of the study; standard clinical care is provided. Data collection focuses on identifying clinical and laboratory predictors of hospitalization and transfusion, including platelet count, hematocrit changes, bleeding signs, and warning symptoms. Transfusion decisions are made independently by the attending physicians, and their rationale is recorded for analysis.

SUMMARY:
This 3-year prospective observational study aims to identify clinical and laboratory risk factors associated with hospitalization in patients with confirmed dengue virus infection. It also seeks to analyze real-world transfusion practices and their outcomes. The study will be conducted in a second-level hospital in northern Mexico and will follow patients from emergency department entry to clinical resolution or hospital discharge.

DETAILED DESCRIPTION:
This study will prospectively follow patients over 3 years to determine the relationship between clinical/laboratory variables and outcomes such as hospitalization and transfusion need. It seeks to improve understanding of real-world decision-making in transfusions for dengue-related thrombocytopenia and refine current hospitalization criteria based on locally observed predictors.

Patients will be enrolled consecutively at emergency departments or outpatient clinics with confirmed dengue infection. Clinical data (fever duration, bleeding signs, vomiting, abdominal pain, platelet count, hematocrit) and transfusion records will be collected and analyzed to identify independent predictors using multivariate logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥5 years
* Laboratory-confirmed dengue infection (NS1, IgM, or PCR)
* First contact at emergency or outpatient services
* Informed consent signed by the patient or legal guardian

Exclusion Criteria:

* Co-infection with other arboviruses or COVID-19
* Pre-existing hematologic or oncologic disease
* Refusal to sign informed consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of patients with confirmed dengue virus infection who seek care at Clínica México, a second-level hospital located in Piedras Negras, Coahuila, Mexico. Participants will be enrolled from both the emergency department and outpatient services. The hospital primarily serves an urban and peri-urban population from northern Coahuila and bordering rural areas. This setting allows for the inclusion of a broad range of clinical presentations, from mild outpatient cases to severe dengue requiring hospitalization or intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-08-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of enrolled patients requiring hospitalization | Time Frame: Within 10 days of symptom onset
  The proportion of patients with laboratory-confirmed dengue infection who require hospitalization will be recorded. Hospitalization is defined as admission to the inpatient ward or intensive care unit for ≥24 hours due to dengue-related clinical indications.
  Unit of Measure:
  Percentage of participants (%)
Clinical and laboratory risk factors associated with hospitalization | Within 10 days of symptom onset
  Description:
  Among patients who are hospitalized, relevant clinical signs (e.g., persistent vomiting, mucosal bleeding, abdominal pain) and laboratory parameters (e.g., platelet count, hematocrit rise, leukopenia) will be analyzed to identify independent predictors for hospitalization using multivariate regression.
  Unit of Measure:
  Odds ratio for each factor (as determined by statistical modeling)

SECONDARY OUTCOMES:
Proportion of patients receiving blood product transfusion | Time Frame: Within 14 days
  The proportion of participants who receive any blood product transfusion (platelets, red cells, plasma) will be documented. Transfusions must be indicated for dengue-related complications and recorded in the patient file.
  Unit of Measure:
  Percentage of participants (%)
Criteria for transfusion used by attending physicians | Within 14 days of symptom onset
  Documented clinical and laboratory criteria used to justify transfusion (e.g., platelet count < 20,000/μL with bleeding, hemodynamic instability, or major hemorrhage) will be analyzed descriptively. No interventions will be assigned by the study team.
  Unit of Measure:
  Proportion of cases using each transfusion criterion (%)

OTHER OUTCOMES:
ICU admission or mortality | Time Frame: 30 days
  Proportion of patients who require intensive care unit admission or who die during the course of illness will be recorded to characterize disease severity.
  Unit of Measure:
  Percentage of participants (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Mexico, Piedras Negras, Coahuila, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided.

REFERENCES:
- [Background] Kalayanarooj S, Vaughn DW, Nimmannitya S, Green S, Suntayakorn S, Kunentrasai N, Viramitrachai W, Ratanachu-eke S, Kiatpolpoj S, Innis BL, Rothman AL, Nisalak A, Ennis FA. Early clinical and laboratory indicators of acute dengue illness. J Infect Dis. 1997 Aug;176(2):313-21. doi: 10.1086/514047. PMID 9237695